CLINICAL TRIAL: NCT01605279
Title: Randomised Double Blind Clinical Trial of Dobutamine Versus Placebo for Low Superior Vena Cava Flow Treatment in Low Birth Weight Infants: Systematic Assessment of Cerebral and Systemic Hemodynamics Effects
Brief Title: Dobutamine Versus Placebo for Low Superior Vena Cava Flow in Newborns
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adelina Pellicer (Other)
Responsible Party: Sponsor-Investigator, Adelina Pellicer, Principal investigator, Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz
Organization: Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NeoDobuta; 2009-010901-35 (EudraCT Number)
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Hemodynamic Instability
Keywords: Low superior vena cava flow; Functional echocardiography
MeSH Terms: interventions — Dobutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dobutamine (Experimental): Patients with low SVCF in the first 12 hours of life will be randomised to receive dobutamine or placebo.
  Interventions: Drug: Dobutamine
- Placebo (Placebo Comparator): Patients with low SVCF in the first 12 hours of life will be randomised to receive Dobutamine or Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dobutamine — Patients with low SVCF in the first 12 hours of life will be randomized to receive Dobutamine or Placebo. First dose: 5 microg/k/min; second dose: 10 microg/k/min; third dose: 15 microg/k/min; forth dose: 20 microg/k/min. Dobutamine concentration will be prepared in a 20 ml syringe and the dose will be adjusted so each 0.1 ml/kg per hour increase in flow rate would deliver the corresponding step-increase in the drug infusion dose. Dose increments will be 5, 10, 15, 20 microg/kg per minute The study drug was increased in a stepwise manner every 30 minutes until the optimal SVCF was attained and maintained for 60 minutes (SVCF-OP). Treatment duration: 24 hours of postnatal age, maintaining the infusion rate which achieves the SVCF-OP.
  Other Names: DB
  Arms: Dobutamine
Drug: Placebo — Patients with low SVCF in the first 12 hours of life will be randomised to receive Dobutamine or Placebo (dextrose 5% in water, D5W, as Placebo)
  Other Names: PL
  Arms: Placebo

SUMMARY:
Low systemic flow as measured by Doppler-echocardiography has been associated with poor neurological outcome. Yet, it has not been systematically evaluated whether the treatment of this hemodynamic condition is beneficial or not. This study aims to evaluate if treating low systemic flow in preterm infants with dobutamine has any effect on the cerebral circulation and in newborn prognosis.

DETAILED DESCRIPTION:
While rates of survival for very preterm infants are increasing, a significant number of these patients suffer from neurodevelopmental disabilities. The pathophysiology of brain injury in the preterm infant is unclear, although haemodynamic disturbances during the period of transitional circulation after birth leading to ischemia-reperfusion events seem to play an important role. Up to one third of infants born under 30 weeks of gestation develop low systemic flow as measured by Doppler-echocardiography (low superior vena cava flow, SVCF); this finding has been associated with poor neurological outcome. Yet, it has not been systematically evaluated whether the treatment of this hemodynamic condition is beneficial or not. This study aims to evaluate if treating low systemic flow in preterm infants with dobutamina, DB, (inotrope-sympathicomimetic drug) has any effect on the cerebral circulation; specific interest of our research would be to target DB dose for individual patient´s response. Secondly, by means of two non-invasive technologies (cerebral and cardiac ultrasonography-Doppler and near infrared spectroscopy, NIRS), the investigators search to characterise eventual differences in brain perfusion patterns during the adaptation to the transitional circulation that might be associated with the development of brain injury in the most vulnerable population.

ELIGIBILITY:
Inclusion criteria

* Newborn infants born at ≤ 28 weeks of gestational age.
* Newborn infants born at > 28 weeks of gestational age and ≤ 30 weeks of gestational age with moderate-severe respiratory distress syndrome, defined as the necessity of respiratory support with a mean pressure ≥ 4 cm H2O or FiO2 ≥ 0.3
* Admission at the NICU in the first 6 hours of life
* Inotrope treatment absent
* Inform consent signed

Exclusion criteria

* Early systemic hypotension, defined as a mean arterial pressure (MAP) lower than the gestational age, during at least 60 minutes and maintained after volume infusion
* Major congenital malformation
* Informed consent declined

Max Age: 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Low SVCF prevalence | From birth to the 4th day of postnatal life
  Low superior vena cava flow (SVCF) prevalence (<40cc/kg/min ) assessed with echocardiography

SECONDARY OUTCOMES:
Required dose for achieving SVCF-OP (≥40 cc/kg/min) | From birth to the 4th day of postnatal life
  Required dose of dobutamine for achieving superior vena cava flow optimum (SVCF-OP) that is SVCF ≥40 cc/kg/min
Required dose for achieving SVCF-OP-60 (≥40 cc/kg/min maintained during 60 minutes) | From birth to the 4th day of postnatal life
  Required dose of dobutamine for achieving superior vena cava flow optimum for 60 min (SVCF-OP-60), that is SVCF ≥40 cc/kg/min maintained during 60 minutes
NIRS variables | From birth to 24 hours of life
  NIRS variables: TOI (tissue oxygenation index), ∆HbT (as a marker of changes in cerebral blood volume, ΔDHb (as a marker of changes in cerebral blood flow will be monitored continuously by NIRS.
Doppler-cranial ultrasonography (PD-CUS) variables. | From birth to the 4th day of postnatal life
  Doppler-cranial ultrasonography (PD-CUS) variables. Changes in cerebral blood flow velocities and the resistance index in cerebral arteries will be evaluated. The effect of SVCF changes on these variables will be analysed.
Invasive or non-invasive arterial blood pressure | From birth to the 4th day of postnatal life
  Invasive or non-invasive arterial blood pressure
Central and peripheral temperature | From birth to the 4th day of postnatal life
  Central and peripheral temperature
Heart rate | From birth to the 4th day of postnatal life
  Heart rate
Respiratory rate | From birth to the 4th day of postnatal life
  Respiratory rate
Other echocardiographic variables | From birth to the 4th day of postnatal life
  * Right and left ventricular output
  * Pulmonary pressure
  * Patent ductus arteriosus
Biochemistry markers | From birth to the 4th day of postnatal life
  * Arterial, venous or capillary gasometry, serum lactate
  * Hemogram, ions, glycemia, creatinine, proteins, Troponine I, N-terminal probrain natriuretic peptide(NT-proBNP)
Structural brain damage markers: | From birth to discharge (approximately around 10-15 weeks)
  * Intraventricular hemorrhage (IVH) grade 1.
  * IVH grade 2.
  * IVH grade 3.
  * Periventricular hemorrhagic infarction.
  * Moderate or severe periventricular echogenicity.
  * Persistent periventricular echogenicity.
  * Cyst periventricular echogenicity.
Mortality and neurodevelopment variables | From birth until 2 years of corrected age
  * Mortality rate
  * Cerebral palsy
  * Neurodevelopmental delay

CONTACTS AND LOCATIONS:
Overall Officials: María Carmen Bravo, PhDMD, Principal Investigator — Fundación Investigación Biomédica HULP
Locations (1):
- La Paz University Hospital, Madrid, Madrid, Spain

REFERENCES:
- [Background] Osborn DA, Evans N, Kluckow M, Bowen JR, Rieger I. Low superior vena cava flow and effect of inotropes on neurodevelopment to 3 years in preterm infants. Pediatrics. 2007 Aug;120(2):372-80. doi: 10.1542/peds.2006-3398. PMID 17671064
- [Derived] Bravo MC, Lopez-Ortego P, Sanchez L, Riera J, Madero R, Cabanas F, Pellicer A. Randomized, Placebo-Controlled Trial of Dobutamine for Low Superior Vena Cava Flow in Infants. J Pediatr. 2015 Sep;167(3):572-8.e1-2. doi: 10.1016/j.jpeds.2015.05.037. Epub 2015 Jun 24. PMID 26116470